CLINICAL TRIAL: NCT00083278
Title: A Phase II Study of MDX-010 in Patients With Stage IV Adenocarcinoma of the Breast
Brief Title: Study of MDX-010 in Stage IV Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: MDX010-12; CA184-015 (Other: BMS)
Record Dates: First submitted 2004-05-17; First posted 2004-05-20 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Breast Cancer; Adenocarcinoma
Keywords: Breast Cancer; Stage IV adenocarcinoma of the breast
MeSH Terms: conditions — Breast Neoplasms; Adenocarcinoma | interventions — Ipilimumab

INTERVENTIONS:
Drug: MDX-010

SUMMARY:
This Phase II study is designed to treat patients who have been diagnosed with Stage IV Breast Cancer, which has progressed despite treatment with primary therapies, including hormonal therapy, chemotherapy, and antibody therapy. Thirty-three patients will be treated with the monoclonal antibody MDX-010. The initial antitumor activity profile of MDX-010 will be determined, as well as identification of the induction of any antitumor immunity following the MDX-010 treatment.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent
* diagnosed with Stage IV adenocarcinoma that has progressed despite previous therapy
* at least 18 years of age
* measurable disease defined by RECIST
* must discontinue any alternative therapy used to treat breast cancer at least 4 weeks prior to enrollment and agree to not use such therapies during the duration of the study (patients may continue to receive tamoxifen, bisphosphate therapy and trastuzumab)
* prior radiation must be completed at least 4 weeks prior to enrollment
* ECOG performance status of 0-2
* Negative pregnancy test
* Screening lab values must be met

Exclusion Criteria:

* must be disease free from other cancers for at least 5 years
* symptomatic or untreated brain metastases
* active or history of autoimmune disease
* active HIV, HTLV, HBV or HCV infection
* concurrent medical condition requiring the use of systemic corticosteroids, must be discontinued at least 4 weeks prior to enrollment
* prior therapy with anti-CTLA-4 antibody
* significant organ compromise, uncontrolled heart, liver, lung, or renal disease or other serious illness
* pregnancy or nursing

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2003-05; Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (14):
- United States (14):
  - Sharp Clinical Oncology Research, San Diego, California
  - Wishard Health Services, Indianapolis, Indiana
  - Section of Hematology/Oncology, Indiana Cancer Pavilion, Indianapolis, Indiana
  - Indiana University, Clarian Health Partners, Indianapolis, Indiana
  - Medical Arts Building, Jeffersonville, Indiana
  - Kansas City Oncology and Hematology Group, Kansas City, Kansas
  - Kansas City Oncology and Hematology Group, Overland Park, Kansas
  - LaGrange, La Grange, Kentucky
  - Norton Healthcare Inc, Loiusville Oncology Clinical Research Program, Louisville, Kentucky
  - Suburban Medical Plaza II, Louisville, Kentucky
  - Audubon Oncology/Hematology, Louisville, Kentucky
  - Kansas City Oncology and Hematology Group, Kansas City, Missouri
  - Kansas City Oncology and Hematology Group, Lee's Summit, Missouri
  - Arlington Cancer Center, Arlington, Texas